CLINICAL TRIAL: NCT02846792
Title: A Phase I/II Clinical Trial of Nivolumab and Plinabulin for Patients With Advanced Stage Non-small Cell Lung Cancer That Have Progressed Through First Line Platinum Doublet Chemotherapy
Brief Title: Nivolumab and Plinabulin in Treating Patients With Stage IIIB-IV, Recurrent, or Metastatic Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Immunotherapy approved for NSCLC in the first line setting
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9602; NCI-2016-01009 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9602 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2016-07-19; First posted 2016-07-27 (Estimated); Results first posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: ALK Gene Translocation; EGFR Activating Mutation; Recurrent Non-Small Cell Lung Carcinoma; ROS1 Gene Translocation; Stage IIIB Non-Small Cell Lung Cancer AJCC v7; Stage IV Non-Small Cell Lung Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; NPI 2358

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (plinabulin, nivolumab) (Experimental): Patients receive plinabulin IV over 30 minutes and nivolumab IV over 60 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab; Drug: Plinabulin

INTERVENTIONS:
Biological: Nivolumab — Given IV
  Other Names: Opdivo
Drug: Plinabulin — Given IV
  Other Names: NPI-2358

SUMMARY:
This phase I/II trial studies the side effects and best dose of plinabulin when given together with nivolumab and to see how well they work in treating patients with stage IIIB-IV non-small cell lung cancer that has come back or spread to other places in the body. Monoclonal antibodies, such as nivolumab, may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as plinabulin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving nivolumab and plinabulin together may work better at treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of the combination of nivolumab and plinabulin. (Phase I)

II. To determine the overall response rate (ORR) of treatment with nivolumab with the addition of plinabulin in the treatment of advanced stage non-small cell lung cancer in the second line setting. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the progression free survival (PFS), disease control rate (DCR), duration of response (DOR) and overall survival (OS) of patients treated with nivolumab in combination with plinabulin.

II. To determine the safety and tolerability of the combination of plinabulin and nivolumab.

TERTIARY OBJECTIVES:

I. Patients who have a pre-treatment and/or post cycle one biopsy will have flow cytometry of their tissue to identify infiltration of immune cells, rates of expression of programmed cell death 1 (PD-1), programmed cell death 2 (PD-2) and programmed cell death 1 ligand 1 (PDL1).

OUTLINE: This is a phase I, dose-escalation study of plinabulin followed by a phase II study.

Patients receive plinabulin intravenously (IV) over 30 minutes and nivolumab IV over 60 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically-documented stage IIIB or stage IV, recurrent, or metastatic non-small cell lung cancer (NSCLC)
* Subjects must have received prior platinum doublet based treatment

  * Up to 2 lines of prior systemic therapy for metastatic disease are permitted
  * Adjuvant chemotherapy or concurrent chemoradiation for early stage disease does not count as prior therapy unless subject progressed within 6 months of completion of regimen
  * Patients with known activating mutations in epidermal growth factor receptor (EGFR), or known translocation in anaplastic lymphoma kinase (ALK) or ROS-1 are eligible provided they have progressed on or were intolerant to Food and Drug Administration (FDA) approved targeted therapy
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Subjects, including those in the dose-escalation portion of the study, must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria; imagining must be within 28 days of trial enrollment

  * Target lesions may be located in a previously irradiated field if there is documented (radiographic) disease progression in that site prior to trial enrollment
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Platelets >= 75,000/dL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 mg/dL x upper limit of normal (ULN) (except subjects with Gilbert syndrome who can have total bilirubin =< 3.0 mg/dL)
* Serum creatinine =< 1.5 mg/dL or creatinine clearance >= 60 mL/min
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 times the upper limit of normal if no liver involvement or =< 5 times the upper limit of normal with liver involvement
* For women of child bearing potential, documented negative pregnancy test within two weeks of study entry and agreement to acceptable birth control throughout the trial starting with the screening visit through 120 days after the last dose of study medication

  * Abstinence is an acceptable method of birth control
* Male subjects with a female partner(s) of child-bearing potential must agree to use acceptable birth control throughout the trial starting with the screening visit through 120 days after the last dose of study medication
* Capability to understand and comply with the protocol requirements as and signed informed consent documents

Exclusion Criteria:

* Systemic anticancer therapy within 21 days of the first dose of study drug

  * All adverse events from prior systemic therapy must have either stabilized or returned to baseline
* Prior treatment with nivolumab or any other PD1/PDL1 checkpoint inhibitor
* Major medical conditions that might affect study participation (e.g. uncontrolled pulmonary, renal, or hepatic dysfunction, uncontrolled serious infection, cardiac disease)
* Significant cardiac history:

  * History of myocardial infarction or ischemic heart disease within 1 year before first study drug administration;
  * Uncontrolled arrhythmia;
  * History of congenital QT prolongation;
  * New York Heart Association class III or IV cardiac disease;
  * Uncontrolled hypertension: blood pressure consistently greater than 150 mm Hg systolic and 100 mm Hg diastolic in spite of antihypertensive medication
* History of hemorrhagic diarrhea, inflammatory bowel disease or active uncontrolled peptic ulcer disease; (concomitant therapy with ranitidine or its equivalent and/or omeprazole or its equivalent is acceptable); history of ileus or other significant gastrointestinal disorder known to predispose to ileus or chronic bowel hypomotility
* Subjects with untreated symptomatic central nervous system (CNS) metastases are excluded

  * Subjects are eligible if symptomatic CNS metastases are treated and subjects have neurologically returned to baseline (except for residual signs and symptoms related to CNS treatment) for at least 7 days prior to first dose of study treatment

    * Subjects must be off corticosteroids for at least 7 days prior to first dose of study treatment
* Subjects with leptomeningeal disease are excluded
* Subjects with planned radiation therapy to a target lesion will be excluded
* Radiation therapy within 14 days of the first dose of study drug
* Subjects who are pregnant or breastfeeding are excluded
* Subjects who are unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee are excluded
* Pulmonary conditions such as sarcoidosis, silicosis, idiopathic pulmonary fibrosis, or hypersensitivity pneumonitis are excluded
* Subject who have active non-infectious pneumonitis
* Subjects who have a diagnosis of immunodeficiency or are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Subjects with any active, known, or suspected autoimmune disease; subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll

  * Subjects with asthma that require intermittent use of bronchodilators, inhaled steroids, or local steroid injections would not be excluded from the study
  * Subjects on chronic systemic steroids for any reason would be excluded from the study; the use of topical steroids is allowable
* Any known additional malignancy (with exception of non-melanoma skin cancer, in-situ breast cancer or a malignancy diagnosed >= 3 years ago and with no evidence of requiring active treatment)
* Patients with known active hepatitis B, or hepatitis C will be excluded
* Patients with risk factors for bowel obstruction or bowel perforation (e.g., acute diverticulitis) will be excluded
* Has any serious or uncontrolled active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Santana-Davila, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seattle Cancer Care Alliance/University of Washington Phase I/II trial open label study enrolled patients at a single site between June 2017 and July 2018.
Pre-assignment Details: Five patients were consented and treated.
Period: Overall Study
Arm/Group | Treatment (Plinabulin, Nivolumab)
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline participant measures are based on total eligible, consented and treated patients.
Arm/Group | Treatment (Plinabulin, Nivolumab)
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 70 [59 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Plinabulin and Nivolumab (Phase I)
Description: Defined as no more than 1 of 6 patients experiencing a dose limiting toxicity, graded according to the National Cancer Institute Common Toxicity Criteria version 4.0.
Time Frame: Up to 28 days
Population: Study terminated (stopped prematurely). Immunotherapy approved for NSCLC in the first line setting.
Arm/Group | Treatment (Plinabulin, Nivolumab)
Number analyzed (Participants) | 0

2. Primary Outcome: Overall Response Rate (Phase II)
Description: Defined as the sum of complete and partial responses for more than 8 weeks according to Response Evaluation Criteria in Solid Tumors version 1.1.
Time Frame: Time between receipt of first study drug until disease progression date, unacceptable toxicity or withdrawal of patient consent, assessed up to 16 months
Population: Study terminated (stopped prematurely). Immunotherapy approved for NSCLC in the first line setting.
Arm/Group | Treatment (Plinabulin, Nivolumab)
Number analyzed (Participants) | 0

3. Secondary Outcome: Disease Control Rate
Description: Defined as the proportion of patients with complete response, partial response, and stable disease for more than 8 weeks according to Response Evaluation Criteria in Solid Tumors version 1.1.
Time Frame: as for outcome 2
Population: Study terminated (stopped prematurely). Immunotherapy approved for NSCLC in the first line setting.
Arm/Group | Treatment (Plinabulin, Nivolumab)
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Response
Description: Will be summarized using descriptive statistics (mean, standard deviation, median, minimum and maximum values).
Time Frame: as for outcome 2
Population: Study terminated (stopped prematurely). Immunotherapy approved for NSCLC in the first line setting.
Arm/Group | Treatment (Plinabulin, Nivolumab)
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: Will be summarized using descriptive statistics (mean, standard deviation, median, minimum and maximum values).
Time Frame: Time between receipt of first study drug until death date or last known alive date, assessed up to 16 months
Population: Study terminated (stopped prematurely). Immunotherapy approved for NSCLC in the first line setting.
Arm/Group | Treatment (Plinabulin, Nivolumab)
Number analyzed (Participants) | 0

6. Secondary Outcome: Toxicity Rates
Description: Overall Percentage and number of patients experiencing grade 3 or higher severity of adverse events, graded using the National Cancer Institute Common Toxicity Criteria version 4.0.
Time Frame: Adverse events collected from the time patient received the first dose of study therapy through 28 days following the last dose of study therapy or the start of a new cancer therapy, whichever occurred first, assessed up to 28 days post therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Plinabulin, Nivolumab)
Number analyzed (Participants) | 5
Participants | 4

7. Secondary Outcome: Progression Free Survival
Description: Assessed using Response Evaluation Criteria in Solid Tumors version 1.1.
Time Frame: as for outcome 2
Population: Study terminated (stopped prematurely). Immunotherapy approved for NSCLC in the first line setting.
Arm/Group | Treatment (Plinabulin, Nivolumab)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected from the time patient received the first dose of study therapy through 28 days following the last dose of study therapy or the start of a new cancer therapy, whichever occurred first, assessed up to 28 days post therapy.
Description: Any adverse events leading to a treatment interruption or dose reduction along with all adverse events that are grade 3 and higher were recorded.
Arm/Group | Treatment (Plinabulin, Nivolumab)
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Plinabulin, Nivolumab) (N=5)
Atrioventricular block (Cardiac disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Prophylactic surgical stabilization of the left femoral head and left proximal tibia due to bone metastases
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Progressive disease
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Plinabulin, Nivolumab) (N=5)
Infusion related reaction (General disorders) | 2 (3)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (2) — Radiation therapy to painful bone metastases
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study terminated (stopped prematurely), due to immunotherapy approved for NSCLC in the first line setting. Participant flow, Baseline Characteristics and Adverse Events recorded for 5 patients treated on study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT02846792/Prot_SAP_000.pdf